CLINICAL TRIAL: NCT03475992
Title: Pilot Clinical Evaluation of a Microwave Imaging System for Early Breast Cancer Detection
Brief Title: Pilot Clinical Study on a Low-power Electromagnetic Wave Breast Imaging Device for Cancer Screening Purposes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MVG Industries SAS (Industry)
Collaborators: HRB Clinical Research Facility Galway (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TN.32.1.17.SATF
Record Dates: First submitted 2018-03-12; First posted 2018-03-23 (Actual); Results first posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer; Breast Cyst
MeSH Terms: conditions — Breast Neoplasms; Breast Cyst

STUDY DESIGN:
Intervention Model Description: The study is performed on 3 groups of patients:
  * Group 1: 15 patients with pre-diagnosed breast cancer (core needle biopsy performed ≥14 days before the microwave breast investigation).
  * Group 2: 10 patients with breast cyst. No prior biopsy
  * Group 3: 5 patients with pre-diagnosed benign lesion (core needle biopsy performed ≥14 days before the microwave breast investigation).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pre-diagnosed breast cancer (Experimental): Low-power microwave breast imaging system.
  Core needle biopsy performed ≥14 days before the microwave breast investigation
  Interventions: Device: Low-power microwave breast imaging system
- Pre-diagnosed breast cyst (Experimental): Low-power microwave breast imaging system.
  No prior biopsy
  Interventions: Device: Low-power microwave breast imaging system
- Pre-diagnosed benign lesion (Experimental): Low-power microwave breast imaging system.
  Core needle biopsy performed ≥14 days before the microwave breast investigation
  Interventions: Device: Low-power microwave breast imaging system

INTERVENTIONS:
Device: Low-power microwave breast imaging system — Investigate the capacity of microwave imaging to detect and characterise diagnosed palpable breast lump

SUMMARY:
The trialed investigational medical imaging device is a low-power microwave breast imaging system for cancer screening purposes. It is an active device which uses non-ionizing radiation.

Microwave imaging is an emerging imaging modality for the early detection of the breast cancer. The physical basis of microwave imaging is the dielectric contrast between healthy and cancerous breast tissues at microwave frequencies. Microwave imaging can potentially be used for monitoring neoadjuvant chemotherapy treatment, breast health monitoring, and for routine screening and diagnosis of the breast cancer at the early-stage. The non-invasive and the non-ionizing characteristics of microwaves should allow for frequent scans of the breast using microwave imaging, unlike X-ray mammography. In addition to safety, microwave imaging does not require uncomfortable breast compression and it is potentially a lower-cost modality.

This is a first-in-human clinical test of the investigational device, which has been so far tested only with experimental phantoms modelling the human female breast.

The clinical data that will be collected in the context of this study is intended to provide early safety information for the investigational medical imaging device. In addition, this exploratory data will guide the refinement of the device hardware and the imaging algorithm design, before decision to proceed (or not) with further clinical tests.

Furthermore, this study will be used to guide sample size calculation for a subsequent study designed to evaluate efficacy should that appear warranted once this study is completed.

DETAILED DESCRIPTION:
This is a single-site early-phase pilot clinical study, taking place at Galway University Hospital/HRB Clinical Research Facility, Galway.

Patients will have a conventional history and breast examinations (Mammogram and / or Ultrasound and Clinical assessment) performed by the physician, as per normal practice in the Symptomatic Breast Unit of University Hospital Galway.

If patients are interested in the study, provide written informed consent and are deemed eligible, they will attend the Clinical Research Facility Galway for a Microwave Breast Imaging (MBI) scan. The data from the scan will be collected and stored securely. Patients will be followed up 7-21 days after the microwave breast investigation or before surgery, whichever comes first. Patients will be assessed for their experience of the microwave breast investigation, and for any adverse events.

The investigational medical imaging device consists of two subsystems, both performing a non-invasive examination:

* the Microwave Breast Imaging subsystem (MBI subsystem);
* the Optical Breast Contour Detection subsystem (OBCD subsystem);

The MBI subsystem is an active device which uses non-ionizing radiation. It illuminates the breast with low-power electromagnetic waves in the microwave frequency spectrum, which penetrate the breast under examination. The subsystem collects the scattered electromagnetic waves and recovers useful information on the breast tissue consistency, given the dielectric contrast of these tissues.

Multi-static radar detection technology is employed in the MBI subsystem for breast image formation.The well-established Microwave Vision Group (MVG) technology for fast antenna measurement, using multiple sensors in a vertical arch configuration, has been transposed to a horizontal arch of sensors. In addition, vertical translation of the horizontal arch has been enabled, such that 3D multi-static short-range radar imaging is possible.

The sensors are in contact with a cylindrical container filled with a liquid; the so-called coupling liquid has been designed to have electromagnetic (EM) properties appropriately selected such that the EM wave penetration in the breast is maximized.

During the MBI scan, the patient is lying in a face down position on a special bed, integrated with the MBI subsystem. The breast under examination is immersed in the coupling liquid, through a dedicated circular opening of the bed. The breast is then scanned. This vertical scan takes approximately 10-15 minutes to complete, depending on the size of each breast.

In order to compute the required volume of coupling liquid, such that the container of the MBI subsystem is optimally filled after immersion of the breast, a simple process for optical assessment of the total volume of the breast takes place just before starting the MBI scan.

The Optical Breast Contour Detection (OBCD) subsystem serves to provide the total volume of the breast, and also its external contour, as a priori information to the MBI subsystem. The OBCD subsystem consists of a 3D optical camera placed below the examination table, at a distance of several tens of centimetres below the breast. An azimuthal scan of the 3D camera permits to reconstruct the external surface of the breast.

In order for the breast contour to be a useful a priori information for the MBI subsystem, it is important that the patient is lying in the same face down position during both the MBI and OBCD scans. Thus, an identical examination table, as the one integrated with the MBI subsystem, is also integrated with the OBCD subsystem. During the OBCD scan, the patient is lying on the examination table, with her breast under examination inserted in the circular opening of the examination table. For this scan, there is no coupling liquid; the breast is in the air, hanging below the examination table.

Both the breast bearing the palpable lump and the contralateral breast will be scanned. The contralateral breast scan will serve as control in the data analysis.

The MBI scan duration of each breast should not exceed 15 minutes. The recorded data will be checked and in the case of non-optimal positioning of the patient, the scan may be repeated.

It is expected that the duration of the microwave breast investigation (including OBCD scan of both breasts for breast volume assessment, preparation of the MBI subsystem, MBI scan of both breasts, and data verification) should not exceed 1 hour. If the Data Quality Check suggests repetition of the MBI scan, and upon agreement by the patient, the total duration of the microwave breast investigation will be extended.

The written radiology reports from conventional imaging will be acquired and used to evaluate the performance of the MBI subsystem in terms of detecting and estimating the size and consistency of the breast lump.

MBI data analysis will be performed off-line, at MVG premises (France), and is expected to be completed few months after the end-date of data collection. Following the assessment of the MBI results by the medical experts involved in the study, a decision will be made regarding the potential of this emerging imaging modality and the interest in proceeding with clinical studies involving larger sample sizes. Based on these results, MVG will decide and plan actions for refinement of the system, towards an upgraded version to be used for potential future tests with a more significant impact.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be able and willing to give written informed consent and to comply with the requirements of this study protocol
2. Subject must have attended the Symptomatic Breast Unit with a palpable breast lump
3. Subjects must have had a mammogram in the clinical assessment period (≤ 6 weeks before the microwave breast investigation)
4. Subjects must be able to comfortably lie reasonably still in a prone position for up to 15 minutes
5. Subjects with bra size larger than 32B and cup size larger or equal to B.
6. Subjects whose breast size is adapted to the cylindrical container of the MBI system with sufficient margin to allow the presence of transition liquid around the breast. Final decision to be taken by the physicians based on their judgement.

Exclusion Criteria:

1. Subjects unable to provide written informed consent
2. Subjects who are pregnant or breast-feeding
3. Subjects who have had previous surgery to the breast
4. Subjects who have previously received chemotherapy or radiotherapy to the breast
5. Subjects who have had a breast biopsy less than two weeks prior to imaging
6. Subjects with any active or metallic implant (e.g. cardiac pacemaker, stents, internal cardiac defibrillator, cardiac resynchronisation device, nerve stimulator…), or subjects bearing any non-removable metallic object (e.g. piercing) on their torso
7. Post-biopsy patients whose breast tissue is not healed sufficiently for the imaging procedure, in the opinion of the investigator
8. Patients who have had or plan to have a breast cyst aspiration before MBI.
9. Subjects with significant co-morbidities which, in the opinion of the investigator, may influence the result of the study
10. Subjects with prior or concurrent malignancy
11. Subjects under the age of 18 years old
12. Subjects with evidence of inflammation and/or erythema of the breast as well as any subjects who have a break in the skin which would be in contact with the coupling fluid
13. Subjects who would be unsuitable for an MBI scan, unlikely to attend a follow up visit, or would otherwise be unsuitable for such an investigation, in the opinion of the Investigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2020-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kerin, Prof., Principal Investigator — Galway University Hospital
Locations (1):
- HRB Clinical Research Facility Galway, Galway, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The manufacturer of the trialed investigational medical device and sponsor of the clinical investigation — http://www.mvg-world.com/en
- See also: The investigational site — http://www.nuigalway.ie/hrb_crfg/

RESULTS

PARTICIPANT FLOW:
Groups:
- Pre-diagnosed Breast Cancer - Biopsy Confirmed; Pre-diagnosed Benign Lesion - Biopsy Confirmed: Low-power microwave breast imaging system.
  Core needle biopsy performed ≥14 days before the microwave breast investigation
  Low-power microwave breast imaging system: Investigate the capacity of microwave imaging to detect and characterise diagnosed palpable breast lump
- Pre-diagnosed Breast Cyst: Low-power microwave breast imaging system.
  No prior biopsy
  Low-power microwave breast imaging system: Investigate the capacity of microwave imaging to detect and characterise diagnosed palpable breast lump
Period: Overall Study
Arm/Group | Pre-diagnosed Breast Cancer - Biopsy Confirmed | Pre-diagnosed Breast Cyst | Pre-diagnosed Benign Lesion - Biopsy Confirmed
Started | 11 | 9 | 5
Completed | 11 | 9 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Overall, there have been twenty-five (25) patients scanned with the low-power Microwave Breast Imaging (MBI) system. Out of the twenty-five (25) patients, twenty-four (24) were included in the final analysis. The patient who was excluded from the final analysis was a patient who presented with a palpable lump which was subsequently determined to be normal breast tissue
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-diagnosed Breast Cancer - Biopsy Confirmed | Pre-diagnosed Breast Cyst | Pre-diagnosed Benign Lesion - Biopsy Confirmed | Total
Number analyzed (Participants) | 11 | 8 | 5 | 24
Age, Continuous [Mean (Full Range); unit: years] | 64.6 [42 to 83] | 38.3 [35 to 49] | 39.4 [36 to 47] | 50.5 [35 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 5 | 24
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Irish | 10 | 7 | 5 | 22
  Race: Brazilian | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Ireland | 11 | 8 | 5 | 24
Volumetric Breast Density [Mean (Full Range); unit: Percentage(%) of dense tissue volume] — Population: The "For processing" DICOM mammography data was unavailable for four (4) of the twenty-four (24) analysed patients due to accidental deletion/retention of data. This data is required to compute the Volumetric Breast Density (VBD) with the Volpara VDM software.
  VBD was computed on both breasts of each patient (total number of samples = 40).
  Percentage(%) of dense tissue volume
    number analyzed (Participants) | 9 | 7 | 4 | 20
    (all) | 8.01 [4.00 to 15.40] | 18.04 [8.40 to 27.40] | 13.22 [5.80 to 25.45] | 12.56 [4.00 to 25.45]
Breast Volume [Mean (Full Range); unit: milliliters (mL)] — Population: The "For processing" DICOM mammography data was unavailable for four (4) of the twenty-four (24) analysed patients due to accidental deletion/retention of data. This data is required to compute the Breast Volume with the Volpara VDM software.
  The volume of both breasts of each patient was computed (total number of samples = 40).
  milliliters (mL)
    number analyzed (Participants) | 9 | 7 | 4 | 20
    (all) | 757.3 [293 to 1369] | 647.8 [150 to 1338] | 646.5 [222.7 to 1105.6] | 696.8 [150 to 1369]

OUTCOME MEASURES:

1. Primary Outcome: Number of Serious Adverse Events, Directly Related to Normal Functioning of the Device
Description: To provide early safety information for the proposed investigational medical imaging device.
Time Frame: Through study completion, up to 21 days
Population: All patients who had a low-power Microwave Breast Imaging (MBI) scan completed
Measure: Number; unit: Serious Adverse Events
Arm/Group | Pre-diagnosed Breast Cancer - Biopsy Confirmed | Pre-diagnosed Breast Cyst | Pre-diagnosed Benign Lesion - Biopsy Confirmed
Number analyzed (Participants) | 11 | 9 | 5
Serious Adverse Events | 0 | 0 | 0

2. Other Pre Specified Outcome: Capacity of the Low-power Microwave Breast Imaging (MBI) System to Detect Pre-diagnosed Palpable Breast Lesions. Detection Rate for Malignant and Benign Breast Lesions.
Description: Percentage of total number of biopsy-confirmed malignant breast lesions being detected with MBI; Percentage of total number of pre-diagnosed breast cysts being detected with MBI; Percentage of total number of biopsy-confirmed benign breast lesions being detected with MBI.
Time Frame: Duration of study - 19 months
Population: as for baseline characteristics
Measure: Number; unit: Percentage(%) of lesions being detected
Arm/Group | Pre-diagnosed Breast Cancer - Biopsy Confirmed | Pre-diagnosed Breast Cyst | Pre-diagnosed Benign Lesion - Biopsy Confirmed
Number analyzed (Participants) | 11 | 8 | 5
Percentage(%) of lesions being detected | 82 | 100 | 80

ADVERSE EVENTS:
Time Frame: Safety data collected over 15 months
Arm/Group | Pre-diagnosed Breast Cancer - Biopsy Confirmed | Pre-diagnosed Breast Cyst | Pre-diagnosed Benign Lesion - Biopsy Confirmed
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9 | 0/5
Other Adverse Events (participants affected / at risk) | 0/11 | 1/9 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-diagnosed Breast Cancer - Biopsy Confirmed (N=11) | Pre-diagnosed Breast Cyst (N=9) | Pre-diagnosed Benign Lesion - Biopsy Confirmed (N=5)
Eyelid infection-stye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — Stye on upper eyelid of patient's right eye

LIMITATIONS AND CAVEATS:
First in Human, exploratory, open clinical study was conducted in order to gather clinical data to support refinement of Prototype # 1 of the low-power MBI system as well as initial safety information

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/92/NCT03475992/Prot_SAP_000.pdf